CLINICAL TRIAL: NCT02534675
Title: An Open Label Navigational Investigation of Molecular Profile-Related Evidence Determining Individualized Cancer Therapy for Patients With Incurable Malignancies and Poor Prognosis
Brief Title: Study of Molecular Profile-Related Evidence to Determine Individualized Therapy for Advanced or Poor Prognosis Cancers
Acronym: I-PREDICT
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Principal Investigator, Jason K. Sicklick, M.D., Assistant Professor, Surgery, University of California, San Diego
Other Study IDs: 141758
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Primary tumor tissue or metastases
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to learn more about personalized cancer therapy including response to treatment and side effects. Information from the patient's medical record regarding the tests and treatments they have received, or will receive, for their cancer will be collected. Genomic testing on tissue from the primary tumor or metastases will be used to match therapy recommendations. Patients in which there is no appropriate matched therapy will receive systemic chemotherapy according to their treating physician's discretion. This information will be used to describe whether or not patients respond better when their physicians choose to treat them according to the genetic makeup of their tumor.

DETAILED DESCRIPTION:
This is a prospective, open label navigational investigation to evaluate the feasibility of using molecular profile-based evidence to determine individualized cancer therapy for patients with incurable malignancies. This is a non-randomized, histology-agnostic trial. While it is known that individual histologies are composed of a heterogeneous mix of genomic alterations, it is not clear that one case mix is better or worse than another. Thus, a strategy of molecular matching that may apply across cancers is being tested. All eligible and consented patients will have their tumor tissues genomic profiled by Foundation Medicine's FoundationOne genomic analysis. Patients will be stratified into Group 1 (treatment naïve, unresectable/medically unfit for surgery), Group 2 (treatment naïve, metastatic), and Group 3 (prior treated), respectively. Following analysis for genomic alterations, matched therapy, if available, will be recommended by the Study Committee or Molecular Tumor Board. If the patients received the matched therapy, they are designated as in Arm A. Otherwise, if the patients received the unmatched therapy (i.e., treating physician's choice of traditional systemic chemotherapy), they are designated as in Arm B. The study feasibility will be measured by the ability to enroll patients, the acceptable turnaround time and the actionable information obtained from the genomic profiling, and the viability of identifying and delivering the matched therapy. The treatment efficacy will be determined among the patients groups and treatment arms. The safety profile of the treatment will also be assessed.

ELIGIBILITY:
Inclusion Criteria Patients must meet all of the inclusion criteria to participate in this study.

1. Patients with incurable malignancies with more than 50% 2-year cancer-associated mortality (as estimated by two physician and where appropriate according to 2014 National Cancer database)

   Diseases include, but are not limited to:

   Ampullary carcinoma Intrahepatic cholangiocarcinoma (IHCC) Appendiceal cancer Melanoma Colorectal cancer (CRC) Non-KIT GIST (gastrointestinal stromal tumor) Extrahepatic cholangiocarcinoma (EHCC) Non-small cell lung cancer (NSCLC) Esophageal adenocarcinoma Ovarian cancer Gallbladder cancer (GBCA) Pancreatic ductal adenocarcinoma (PDAC) Gastric adenocarcinoma Sarcoma (high-grade) Head and neck cancer Small bowel adenocarcinoma (including duodenal) Hepatocellular carcinoma (HCC) Triple-negative breast cancer (TNBC) Urothelial cancer
2. Patients with cancer of unknown primary or a rare tumor (for example, fewer than 15 cases per 100,000 per year) with no approved therapies. (Patients in this inclusion criteria must meet all other exclusion and inclusion criteria except inclusion criteria #1)
3. Patients with incurable malignancies, irrespective of 2-year mortality, who, in the opinion of the investigator have no treatment option expected to yield significant clinical benefit."
4. Patients must have at least one of the following for a diagnosis/disease status:

   1. Unresectable disease
   2. Metastatic disease
   3. Medically unfit for surgical resection but with an expected survival of > 3 months, ECOG < 2 and NYHA status ≤ II (refer to status definitions in tables below)
   4. Disease where no conventional therapy leads to a survival benefit > 6 months in the respective cohort and line of therapy for which the patient is otherwise eligible
   5. Actionable alterations determined by FoundationOneTM
5. Treatment naïve for his or her newly diagnosed malignancy for enrollment to Groups 1 or 2.
6. Status post 1 or more unmatched systemic therapy regimens for enrollment to Group 3.
7. Ability to understand and the willingness to sign a written informed consent.
8. Patients must have measurable disease for malignancies: defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, PET-CT, MRI, or calipers by clinical exam.
9. Age ≥ 18 years.
10. ECOG Performance Status 0-1.

    Grade Description 0 Fully active, able to carry on all pre-disease performance without restriction 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework or office work 2 Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours 3 Capable of only limited self-care, confined to a bed or chair >50% of waking hours 4 Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair 5 Dead
11. New York Heart Association (NYHA) Functional Classification I-II.

    NYHA Class Symptoms I Cardiac disease, but no symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.

    II Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.

    III Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).

    Comfortable only at rest. IV Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
12. Adequate organ and marrow function as defined below:

    * Absolute neutrophil count ≥ 1.5 x 109/L
    * Platelet count ≥ 100 x 109/L
    * Total bilirubin ≤ 2.0 x institution's ULN
    * Patients without underlying liver disease

      o ALT and AST ≤ 2.5 X institutional upper limit of normal
    * Serum creatinine ≤ 2.0 x institution's ULN or 24-hour creatinine clearance ≥ 50 ml/min
13. At the time of treatment, patients should be off other anti-tumor agents for at least 5 half-lives of the agent or 3 weeks from the last day of treatment, whichever is shorter to enroll in Group 3. Patients must not have been treated with anti-tumor agents to enroll in Group 1 or Group 2. Patients must be off prior antibody therapy for at least 3 half-lives before starting treatment. Patients may enroll on study even while receiving treatment.
14. Able to swallow and retain oral medication if needed.
15. Patients must have evaluable tissue/blood for testing as specified by the concurrent FoundationOneTM criteria. This will be obtained during the standard of care tumor diagnosis and tumor staging evaluation.
16. Female patients of childbearing potential must have a negative serum pregnancy test and agree to use at least one form of pregnancy prevention during the study and for at least one month after treatment discontinuation. For the purposes of this study, child- bearing potential is defined as: all female patients that were not in post- menopause for at least one year or are surgically sterile (site-specific criteria applying to Avera only)
17. Male patients must use a form of barrier pregnancy prevention approved by the investigator / treating physician during the study and for at least one month after treatment discontinuation (site-specific criteria applying to Avera only).

Exclusion Criteria Subjects meeting any of the exclusion criteria at baseline will be excluded from study participation.

1. Two oncologists disagree on prognosis or resectability.
2. Severe or uncontrolled medical disorder that would, in the investigator's opinion, confound study analyses of treatment response (i.e., uncontrolled diabetes, chronic renal disease, chronic pulmonary disease or active, uncontrolled infection, psychiatric illness/social situations that would limit compliance with study requirements).
3. Are pregnant or breast-feeding patients or any patient with childbearing potential not using adequate pregnancy prevention (site-specific criteria applying to Avera only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with incurable malignancies with aggressive biology
Sampling Method: Non-Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2015-02; Primary Completion 2020-12-17 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who receive the molecularly targeted matched treatment after recommendations based on genomic analysis | 3 years
  Number of patients who received study therapy after recommendations after genetic test versus patients who did not

SECONDARY OUTCOMES:
Proportion of patients who consent to enroll into the study | 3 years
  To calculate the number of patients who have consented to be on the study
Time from informed consent to receipt of genomic analysis | 3 years
  To calculate the time between getting the patient's consent and them receiving their genetic test
Proportion of patients with actionable genomic alteration | 3 years
  To calculate the number of patients who have a genetic test result that can be matched with appropriate treatment that can target their specific mutation
Proportion of patients with insurance coverage for receiving molecularly targeted matched treatment based on genomic analysis | 3 years
  To calculate the number of patients who are covered by insurance to receive treatment appropriately targeting their specific genetic test result

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sicklick, MD and Razelle Kurzrock, MD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - UCSD Moores Cancer Center, La Jolla, California
  - Avera Cancer Institute, Sioux Falls, South Dakota

REFERENCES:
- [Derived] Noh S, Sharma AK, Fanta PT, Kato S, Kurzrock R, Sicklick JK. Personalized N-of-1 Combination Therapies for Advanced Gastrointestinal Stromal Tumors. JCO Precis Oncol. 2025 Jul;9:e2500066. doi: 10.1200/PO-25-00066. Epub 2025 Jul 23. PMID 40700673
- [Derived] Sicklick JK, Kato S, Okamura R, Patel H, Nikanjam M, Fanta PT, Hahn ME, De P, Williams C, Guido J, Solomon BM, McKay RR, Krie A, Boles SG, Ross JS, Lee JJ, Leyland-Jones B, Lippman SM, Kurzrock R. Molecular profiling of advanced malignancies guides first-line N-of-1 treatments in the I-PREDICT treatment-naive study. Genome Med. 2021 Oct 4;13(1):155. doi: 10.1186/s13073-021-00969-w. PMID 34607609